CLINICAL TRIAL: NCT01221987
Title: A Cross-sectional, Hospital-based, Epidemiological Study on Human Papillomavirus Type Distribution in Adult Women Diagnosed With Invasive Cervical Cancer (ICC) and/or Cervical Intraepithelial Neoplasia (CIN) II and/or CIN III in Sri Lanka
Brief Title: Cross-sectional Study on Human Papillomavirus Type Distribution in Adult Women Diagnosed With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 110430
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2011-05

CONDITIONS: Neoplasms, Uterine Cervix; Cervical Cancer
Keywords: Human papillomavirus; neoplasia
MeSH Terms: conditions — Neoplasms; Uterine Cervical Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue samples of invasive cervical cancer

GROUPS / COHORTS (2):
- Cohort A: Females > 21 years of age, diagnosed with invasive cervical cancer
  Interventions: Procedure: Cervical sampling; Other: Data collection
- Cohort B: Females > 21 years of age, diagnosed with moderate or severe cervical intraepithelial neoplasia
  Interventions: Procedure: Cervical sampling; Other: Data collection

INTERVENTIONS:
Procedure: Cervical sampling — Cervical biopsy or excision specimen testing for human papillomavirus deoxyribose nucleic acid types
Other: Data collection — Questionnaire completion

SUMMARY:
The current study will elucidate the human papillomavirus type distribution in a population of women diagnosed with cervical high grade pre-cancerous lesions and invasive cervical cancer in Sri Lanka.

ELIGIBILITY:
Inclusion Criteria:

* A female > 21 years of age at the time of diagnosis of invasive cervical cancer or cervical intraepithelial neoplasia - moderate or severe.
* Histologically confirmed diagnosis of cervix intraepithelial neoplasia - moderate or severe, invasive cervical cancer, glandular lesions and other epithelial tumours.
* Written informed consent obtained from the subject prior to study start.
* Subjects who the investigator believes can and will comply with the requirements of the protocol, should be enrolled in the study.

Exclusion Criteria:

* Previous vaccination against human papillomavirus.
* History of chemotherapy or radiotherapy for cervical cancer.
* Subjects with recurrent episodes of invasive cervical cancer or cervical intraepithelial neoplasia- moderate or severe.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females > 21 years of age, diagnosed with invasive cervical cancer or cervical intraepithelial neoplasia - moderate or severe
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Detection of human papillomavirus-16, human papillomavirus-18 in invasive cervical cancer and cervix intraepithelial neoplasia- moderate or cervix intraepithelial neoplasia- severe by short PCR fragment polymerase chain reaction and line probe assay | Up to 12 months from the date of study initiation

SECONDARY OUTCOMES:
Detection of other high risk types in invasive cervical cancer and cervical intraepithelial neoplasia moderate or severe by short PCR fragment polymerase chain reaction and line probe assay | Up to 12 months from the date of study initiation
Occurrence of human papillomavirus-16, human papillomavirus-18 or other high risk types in relation to covariates | Up to 12 months from the date of study initiation
Detection of co-infection of human papillomavirus-16 and human papillomavirus-18 in relation to other high risk types | Up to 12 months from the date of study initiation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Karunaratne K, Ihalagama H, Rohitha S, Molijn A, Gopala K, Schmidt JE, Chen J, Datta S, Mehta S. Human papillomavirus prevalence and type-distribution in women with cervical lesions: a cross-sectional study in Sri Lanka. BMC Cancer. 2014 Feb 21;14:116. doi: 10.1186/1471-2407-14-116. PMID 24558979